CLINICAL TRIAL: NCT00582231
Title: Penile Injection Anxiety
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 07-001
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Penile Injection Therapy; Erectile Dysfunction; Radical Pelvic Surgery
Keywords: Penile injection therapy; Erectile dysfunction; Radical pelvic surgery; Penile Injection Anxiety
MeSH Terms: conditions — Erectile Dysfunction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Participants that are starting penile injections therapy.
  Interventions: Other: Questionnaires.

INTERVENTIONS:
Other: Questionnaires. — Questionnaires.

SUMMARY:
The purpose of this study is to help us understand more about your experience with penile injection therapy. Many men become anxious when thinking about penile injections. We would like to understand more about this anxiety. You will be asked to fill out questionnaires before you start penile injection training, at each training visit, and then at your four month follow-up visit.

DETAILED DESCRIPTION:
The treatment of erectile dysfunction (ED) following radical pelvic surgery has become an increasingly important issue. For many men, oral medications for ED will not be effective immediately postoperatively. These medications enhance the effect of nitric oxide secreted from the cavernous nerves, however these nerves are usually transiently injured intraoperatively diminishing the amount of nitric oxide available. Consequently, oral medications are usually ineffective for up to 18 to 24 months postoperatively while the cavernous nerves are healing. As a result, penile injection therapy is the primary treatment for ED for those men. This treatment delivers intracavernosal vasodilators at the base of the penis with a 29 gauge needle. This direct application produces consistent results and has been found to be effective for 94% of injection users. Despite common sense and clinical experience that indicates men become very anxious about penile injection therapy, anxiety has rarely been assessed in studies of penile injection therapy. We have observed that men who are initially reluctant about penile injection therapy are more likely to try this treatment when they hear that the injection anxiety dissipates quickly, after only a few injections. We unfortunately only have clinical observation to support our claim describing the course of injection anxiety. This study would provide empirical data to support this claim and this data will be used in describing the treatment and encouraging men to try injection therapy.

ELIGIBILITY:
Inclusion Criteria:

* History of a radical pelvic surgery (cystectomy, prostatectomy, low anterior resection)
* Participating in the injection therapy program
* Ability to provide informed consent
* Ability to converse, write and read English

Exclusion Criteria:

* History of or currently receiving radiation therapy,
* History of or currently receiving chemotherapy,
* History of or currently receiving hormone therapy.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants that are starting penile injections therapy.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2007-02; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The general paradigm for assessing outcomes of the trial will be repeated measures analysis of variance (ANOVA) and mixed effects models. To assess the change of anxiety levels in men utilizing penile injection therapy following radical pelvic surgery. | Participants will be asked to complete questionnaires before the start of the penile injection training, at each training visit, and then again at the four month follow-up visit.

SECONDARY OUTCOMES:
To study the effects of penile injection therapy on the related domains of erectile dysfunction (IIEF), relationship satisfaction (RAS), sexual satisfaction (SEAR), and depression (HADS-D). | Participants will be asked to complete questionnaires before the start of the penile injection training, at each training visit, and then again at the four month follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Nelson, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org